CLINICAL TRIAL: NCT03492762
Title: PET Imaging CCR2 in Lung Inflammation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20171192; R01HL151685-01A1 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Lung Inflammation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: 2 groups: Healthy Volunteers and Volunteers with Documented ILD Diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteer Group (Experimental): The healthy volunteer group will receive the same interventions as the ILD documented diagnosed volunteer group
  Interventions: Drug: Cu-DOTA-ECL1i
- ILD Documented Diagnosed Volunteer Group (Experimental): The ILD documented diagnosed volunteer group will receive the same interventions as the healthy volunteer group
  Interventions: Drug: Cu-DOTA-ECL1i

INTERVENTIONS:
Drug: Cu-DOTA-ECL1i — Radiolabeled probe called Cu-DOTA-ECL1i that recognizes CCR2 and propose to image CCR2 in the lung to ultimately guide diagnosis and therapy.

SUMMARY:
The primary objective of this study is to assess the lung distribution of the Positron Emission Tomography (PET) imaging radiotracer Cu-DOTA-ECL1i, which binds to the specific population inflammatory cells, in patients with fibrotic lung diseases. This objective includes sub-studies to assess radiotracer distribution in the lung, the reproducibility of PET scans and the relationship of the scan to distribution of inflammatory cells in human lung tissue. The overall goal is to assess the potential of the radiotracer to track inflammatory cells in lung diseases.

DETAILED DESCRIPTION:
This is a single site, pilot Phase 0/1 clinical trial to establish the uptake of Cu-DOTA-ECL1i in additional patients with ILD fibrotic lung disease (n=60). Healthy volunteers without known pulmonary disease will be recruited as controls (N=5). All subjects will be recruited and undergo one dynamic PET/CT scan to characterize the lung uptake of Cu-DOTA-ECL1i. Among those with pulmonary fibrosis imaging, an arterial catheter will be placed for blood draws in n=10 subjects, an additional sub group of subjects (n=10) will undergo a second PET/CT within two months. A third subgroup of subjects (n=10) who undergo lung transplant will have analysis of CCR2+ cells in their explanted lungs.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 21 years of age or older who have never smoked or current smokers who smoked at least 10 cigarettes per day (1/2 pack) and have smoked at least 100 cigarettes (5 packs) over the past month.
* Screening FEV1 and FVC > 80% of predicted
* Capable of lying still and supine within the PET/CT and PET/MR scanner for ~1 hour and follow instructions for breathing protocol during the CT portion
* No illicit drug use or other inhaled drug use (including pharmacologic agents, recreational agents, or illicit drugs) within the past year
* No known history of cardiac, pulmonary, hepatic or renal disease or diabetes
* No history of claustrophobia or other preventing condition that has previously or would interfere with completion of protocol specified imaging sessions
* Able to comprehend and willing to follow instructions for the study procedures as called for by the protocol
* BMI ≤ 35

Exclusion Criteria:

* Currently enrolled in another study using an investigational drug
* Pregnancy (confirmed by urine pregnancy test)
* Active symptoms or history of cardiac, pulmonary, hepatic or renal disease or diabetes
* Currently taking any prescription medications
* Presence of an implanted device that is incompatible with CT or MRI scanning
* Creatinine > 1.30 mg/dL, AST > 50 Units/L, ALT > 55 Units/L, or total bilirubin > 1.2 mg/dL

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of uptake of Cu-DOTA-ECL1i to lung fibrosis | Through study completion
  To establish the relation of lung uptake of Cu-DOTA-ECL1i compared to fibrosis determined by high resolution chest Computed tomography (CT) scan and clinical status
Change of Cu-DOTA-ECL1i as measured by Positron emission tomography (PET) imaging of lung Standard uptake value (SUV) and Distribution Volume Ratio (DVR) over two months | Through study completion
  Determine reproducibility of Cu-DOTA-ECL1i as measured by Positron emission tomography (PET) imaging of lung Standard uptake value (SUV) and Distribution Volume Ratio (DVR) over two months.
Determine rate of kinetics of Cu-DOTA-ECL1i | Through study completion
  Determine rate of kinetics of Cu-DOTA-ECL1i in circulation of blood at 0-60 min post-injection of Cu-DOTA-ECL1i by analysis of the arterial blood metabolites compared to lung uptake by Positron emission tomography/Computed tomography (PET/CT) imaging

SECONDARY OUTCOMES:
Determine relationship between Cu-DOTA-ECL1i lung tissue as seen by Positron emission tomography (PET) imaging and lung tissue showing C-C Motif Chemokine Receptor 2 (CCR2+) cells | Through study completion
  Determine relationship between Cu-DOTA-ECL1i lung tissue as seen by Positron emission tomography (PET) imaging and lung tissue showing C-C Motif Chemokine Receptor 2 (CCR2+) cells using pulmonary function measures

CONTACTS AND LOCATIONS:
Overall Officials: Steven Brody, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
DE-identified individual participant data for all primary and secondary outcome measures will be made available upon publication of trial results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 1 year of the study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Brody SL, Gunsten SP, Luehmann HP, Sultan DH, Hoelscher M, Heo GS, Pan J, Koenitzer JR, Lee EC, Huang T, Mpoy C, Guo S, Laforest R, Salter A, Russell TD, Shifren A, Combadiere C, Lavine KJ, Kreisel D, Humphreys BD, Rogers BE, Gierada DS, Byers DE, Gropler RJ, Chen DL, Atkinson JJ, Liu Y. Chemokine Receptor 2-targeted Molecular Imaging in Pulmonary Fibrosis. A Clinical Trial. Am J Respir Crit Care Med. 2021 Jan 1;203(1):78-89. doi: 10.1164/rccm.202004-1132OC. PMID 32673071